CLINICAL TRIAL: NCT00152737
Title: Effet Des Gestes de Revascularisation à l'étage Proximal
Brief Title: Objective Evaluation of Proximal Ischemia
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Sanofi-Synthelabo (Industry); Société Française de Médecine Vasculaire (Unknown)
Responsible Party: Sponsor
Other Study IDs: PHRC 03-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Intermittent Claudication; Peripheral Vascular Diseases
Keywords: Intermittent Claudication; Peripheral Vascular Diseases; Blood Gas Monitoring, Transcutaneous; Surgery
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Exercise test with Transcutaneous oxygene pressure — Ce marked devices
Procedure: Ankle and arm pressure values — one test before and one test after surgery

SUMMARY:
The whole study is divided in 4 parallel protocols. The first protocol estimates the reliability of the technique through test-retest recordings. The second protocol aims to prove that exercise Tcpo2 is efficient to estimate the benefit of proximal revascularisation on proximal and distal ischemia in patients suffering stage two lower extremity arterial disease. The third protocol aims at estimating with exercise tcpo2 the eventual apparison of proximal ischemia after aorto-bi-femoral bypasses. The last protocol is a transversal study of patients with aorto-bi-femoral bypasses aiming to analyse the presence of proximal and distal symptoms and ischemia.

The hypothesis for protocol 2 is that TcpO2 at exercise is significantly improved after surgery at the aortic and primary iliac artery. The hypothesis for protocols 3 and 4 relates on the hypothesis that a significant number of patients benefiting aorto-bi-femoral bypass suffer isolated proximal pain/ischemia after surgery.

Amendement to the project has been recently validated to study the neurologic and bone complication of chronic vascular ischemia

DETAILED DESCRIPTION:
Patients included are submitted to:

San Diego Claudication Questionnaire before and during the treadmill test Treadmill test(s) through the Strandness procedure (2MPh 10% slope) Transcutaneous oxygen pressure recording before during and after exercise Ankle and brachial pressure measurements. Neurologic investigation with Quantitative sensory Testing (QST) and neurophysiological tests for patients included in the sub-group analysing neurologic complication Whole body densitometry for patients included in the sub-group analysing osteo-articular complications

ELIGIBILITY:
Inclusion Criteria:

* protocol 1 - 3 stage 2 claudication
* Protocols 2 & 3 : Indication for surgery
* protocol 4 : Patent aorto bio femoral bypass for more than 4 months
* Ability to perform a treadmill test

Exclusion Criteria:

* Stage 4 LEAD
* Aortic aneurysm
* Acute coronary syndrom
* claudication of documented non vascular origin (for protocols 1-3 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with claudication
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2004-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: jean louis Saumet, MD PhD, Study Chair — University Hospital in Angers; Pierre Abraham, MD PhD, Principal Investigator — University Hospital in Angers; Bernard Enon, MD, Study Chair — University Hospital in Angers
Locations (1):
- Laboratoire d'explorations vasculaires, Angers, France

REFERENCES:
- [Result] Jaquinandi V, Picquet J, Bouye P, Saumet JL, Leftheriotis G, Abraham P. High prevalence of proximal claudication among patients with patent aortobifemoral bypasses. J Vasc Surg. 2007 Feb;45(2):312-8. doi: 10.1016/j.jvs.2006.09.050. PMID 17264010
- [Result] Jaquinandi V, Abraham P, Picquet J, Paisant-Thouveny F, Leftheriotis G, Saumet JL. Estimation of the functional role of arterial pathways to the buttock circulation during treadmill walking in patients with claudication. J Appl Physiol (1985). 2007 Mar;102(3):1105-12. doi: 10.1152/japplphysiol.00912.2006. Epub 2006 Nov 16. PMID 17110509
- [Derived] Ouedraogo N, Feuilloy M, Mahe G, Leftheriotis G, Saumet JL, Abraham P. Chest tcpO2 changes during constant-load treadmill walking tests in patients with claudication. Physiol Meas. 2011 Feb;32(2):181-94. doi: 10.1088/0967-3334/32/2/003. Epub 2010 Dec 22. PMID 21178246